CLINICAL TRIAL: NCT02765581
Title: Evaluating the Prophylactic Efficacy of Acupuncture for Migraine Without Aura (MWoA) : A Randomized Controlled Trial
Brief Title: Efficacy Study of Acupuncture in the Prevention of Migraine Without Aura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Wang (Other)
Collaborators: Hubei College of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other); University Hospital of Huang Jia Lake Campus, Hubei University of Chinese Medicine (Unknown); The Second Hospital of Huangshi (Unknown); Xiangyang No.1 People's Hospital, Hubei University of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Wei Wang, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201403RCTMWA
Record Dates: First submitted 2016-04-10; First posted 2016-05-06 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Migraine Without Aura
Keywords: Acupuncture; Migraine without aura; Efficacy; Randomized controlled trial; Non-penetrating sham acupuncture
MeSH Terms: conditions — Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum acupuncture (VA) (Experimental): Participants will be treated by verum acupuncture and usual care. They will be treated every other day to fulfill a 10-session treatment course, and another course will begin after resting 9 days. Each acupuncture treatment session for patients will be 30 minutes in duration.
  Interventions: Device: Verum acupuncture; Behavioral: Usual care
- Sham acupuncture (SA) (Sham Comparator): Participants will be treated by sham acupuncture and usual care. They will be treated every other day to fulfill a 10-session treatment course, and another course will begin after resting 9 days. Each acupuncture treatment session for patients will be 30 minutes in duration.
  Interventions: Device: Sham acupuncture; Behavioral: Usual care
- Usual care (UA) (Placebo Comparator): Participants will undergo a clinical interview once a month, complete the headache diary assessment, have counseling and health education, and rescue medication if necessary. In addition, they will be scheduled to receive 20 sessions of verum acupuncture treatments for free after a waiting period of 24 weeks.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Device: Verum acupuncture — The main acupuncture points are bilateral "Hegu" (L14) and "Taichong" (LR3), unilateral "Taiyang"(EX-HN5), "Fengchi" (GB20) and "Shuaigu" (GB8). Additional points can be chosen according to individual syndrome differentiation of meridians: (1) Yangming headache: Touwei (ST8); (2) Taiyang headache: Tianzhu (BL10); (3) Jueying: Baihui" (GV20). The NO.16 special type of acupuncture (0.30 x 30 mm) produced by German asia-med company will be applied.The needles will be inserted into the skin of acupuncture points and manipulated manually by using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation known as deqi.
  Arms: Verum acupuncture (VA)
Device: Sham acupuncture — We use a non-insertive sham control produced by Asia-med Company in Germany-the streitberger placebo-needle. Sham points are described as follows: 1) Bilateral of midpoint between acupoint "Jianjin"(GB21) and "Jugu"(LI16); 2) 5 cun lateral to the seventh thoracic spine; 3) 5 cun lateral to the eighth thoracic spine; 4) 5 cun lateral to the ninth thoracic spine. Cun is a distance measure unit used in locating acupoints in traditional Chinese medicine (TCM) acupuncture, and the width of patient's thumb interphalangeal joint is regarded as one cun.
  Arms: Sham acupuncture (SA)
Behavioral: Usual care — Health education is provided in three aspects: lifestyle changes, behavioral therapies and migraine self-management.

SUMMARY:
Acupuncture is commonly used for the prevention of migraine, while the evidence for its efficacy is still uncertain. Current studies have not been able to determine whether the efficacy of acupuncture is due to the actual therapeutic effect of acupuncture, or a result of psychological benefits. To address this issue, we designed a clinical trial to evaluate the prophylactic efficacy of acupuncture for migraine without aura (MWoA). Furthermore, we will evaluate the impact of Chinese medicine factors and psychological factors on the efficacy of acupuncture.

DETAILED DESCRIPTION:
This is a multicentre, stratified, randomized, sham-controlled clinical trial. 150 eligible participants will be randomly allocated into verum acupuncture, sham acupuncture, or usual care groups, in a 2:2:1 ratio. The verum acupuncture group will receive twenty verum acupuncture treatments over an eight-week period, while the sham acupuncture group will receive sham acupuncture treatments with non-penetrating needling. Participants assigned to the usual care group are scheduled to receive twenty verum acupuncture treatments for free after waiting 24 weeks. Health education will be provided to participants in the three groups. The primary outcomes will be the changes in the mean number of migraine days and migraine attacks per four-week cycle. The secondary outcomes will be as follows: the proportion of responders, migraine intensity, migraine disability assessment questionnaire, health-related and sleep-related quality of life, the dose of intake of acute medication. Chinese medicine factors will include de qi sensations and Traditional Chinese Medicine (TCM) constitution. Psychological outcomes will include anxiety, depression, personality, expectancy about acupuncture, and doctor-patient relationship. The central randomization and data collection will be conducted by an electronic data management system.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as migraine without aura according to the International Classification of Headache Disorders,3rd edition beta version (ICHD-3β);
2. Aged between 15 and 65 years old, with initial onset of migraines before the age of 50 years; and
3. Experienced migraine attacks for at least 1 year; and
4. Experienced migraine attacks with 2-8 times per month during the last 3 months and baseline period, and the duration of migraine attacks lasting 4-72h without intake of acute drugs or at least 2h with intake of acute drugs; and
5. the mean headache Visual Analogue Scale (VAS) scores 4-8 at baseline; and
6. Had not taken any acupuncture treatment before study entry; and
7. Able to complete the baseline headache diary; and
8. Able to signing a informed consent.

Exclusion Criteria:

1. Tension-type headache, cluster headache, and other primary headache disorders, secondary headache disorders, neuralgia of the face or head; and
2. Combined with cardiovascular, liver, kidney, gastrointestinal tract, blood system and other serious primary diseases affecting the implementation of treatment programs, or combined with epilepsy, Parkinson or other nervous system diseases; and
3. Patients with severe mental illness, such as severe anxiety and depression; and
4. Pregnant women, women in lactation, and those planning to become pregnant; and
5. Participation in other clinical trials; and
6. Illiterate, or patients unable to read and understand scales;
7. Have experience of acupuncture.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change in the number of migraine days | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the mean number of migraine days per 4-week cycle
Change in the frequency of migraine attacks | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the mean number of migraine attacks per 4-week cycle

SECONDARY OUTCOMES:
The proportion of responders | At weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The proportion of patients with at least a 50% reduction of the number of migraine days
Change in visual analogue scale | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the mean visual analogue scale scores per 4-week cycle
Change in Short-Form McGill Pain Questionnaire 2 (SF-MPQ-2). | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the scores of Short-Form McGill Pain Questionnaire 2 (SF-MPQ-2) per 4-week cycle
Change in Migraine Disability Assessment questionnaire(MIDAS). | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.
  The changes in the scores of Migraine Disability Assessment questionnaire(MIDAS)
Change in Migraine-Specific Quality of Life Questionnaire(MSQ) Version 2.1. | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the scores of Migraine-Specific Quality of Life Questionnaire(MSQ) per 4-week cycle
Change in 36-Item Short-Form Health Survey(SF-36). | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the scores of 36-Item Short-Form Health Survey(SF-36) per 4-week cycle
Change in Pittsburgh Sleep Quality Index(PSQI). | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the scores of Pittsburgh Sleep Quality Index(PSQI) per 4-week cycle
Change in the dose of intake of acute medication. | At baseline (four weeks before randomization), weeks 1-4 after randomization, weeks 5-8 after randomization, weeks 9-12 after randomization, weeks 13-16 after randomization, and weeks 17-20 after randomization.
  The changes in the dose of intake of acute medication per 4-week cycle

OTHER OUTCOMES:
The Chinese Version of the Massachusetts General Hospital Acupuncture Sensation Scale | Immediately following each session of acupuncture treatment.
  Acupuncture sensations will be measured by the Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS)
Change in Beck Anxiety Inventory(BAI). | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.
Change in Beck Depression Inventory II(BDI- II). | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.
60-item NEO Personality Inventory-Short Form (NEO-FFI) | At baseline (four weeks before randomization) only once.
Chinese medicine constitution classification | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.
  Patients' Chinese medicine constitution classification will be measured by the score obtained from Constitution in Chinese Medicine Questionnaire (CCMQ)
Acupuncture Expectancy Scale | Before treatment, after the third session of treatment, and after the twentieth session of treatment.
Change in Patient-Doctor Relationship Questionnaire(PDRQ-9) . | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.
Change in Difficult Doctor-Patient Relationship Questionnaire(DDPRQ-10). | At baseline (four weeks before randomization), weeks 5-8 after randomization and weeks 17-20 after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu S, Yu L, Luo X, Wang M, Chen G, Zhang Q, Liu W, Zhou Z, Song J, Jing H, Huang G, Liang F, Wang H, Wang W. Manual acupuncture versus sham acupuncture and usual care for prophylaxis of episodic migraine without aura: multicentre, randomised clinical trial. BMJ. 2020 Mar 25;368:m697. doi: 10.1136/bmj.m697. PMID 32213509